CLINICAL TRIAL: NCT01987752
Title: Safety and Efficacy of Combigan® Ophthalmic Solution in Korea
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: 190342-040
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Results first posted 2014-04-04 (Estimated); Last update posted 2014-04-04 (Estimated); Status verified 2014-02

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Brimonidine Tartrate; Brimonidine Tartrate, Timolol Maleate Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Combigan® Ophthalmic Solution: Patients treated with Combigan® Ophthalmic Solution as per local standard of care in clinical practice.
  Interventions: Drug: brimonidine tartrate/timolol maleate Ophthalmic Solution

INTERVENTIONS:
Drug: brimonidine tartrate/timolol maleate Ophthalmic Solution — brimonidine tartrate/timolol maleate (Combigan®) Ophthalmic Solution as per local standard of care in clinical practice.
  Other Names: Combigan®

SUMMARY:
This study is a Post-Marketing Surveillance study in Korea to evaluate the safety and efficacy of Combigan® (brimonidine tartrate/timolol maleate) Ophthalmic Solution in patients with Open Angle Glaucoma or Ocular hypertension with insufficient response to local beta blockers treated as per standard of care in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Open Angle Glaucoma or Ocular Hypertension treated with Combigan® Ophthalmic Solution as standard of care in clinical practice.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Open Angle Glaucoma or Ocular Hypertension treated with Combigan® Ophthalmic Solution in Clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 732 (Actual)
Dates: Start 2009-01; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Combigan® Ophthalmic Solution
Started | 732
Completed | 732
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combigan® Ophthalmic Solution
Number analyzed (Participants) | 732
Age, Customized [Number; unit: Participants]
  < 50 years | 140
  50 - 59 years | 144
  60 - 69 years | 219
  ≥ 70 years | 225
  Missing Data | 4
Sex/Gender, Customized [Number; unit: Participants]
  Female | 347
  Male | 384
  Missing Data | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Adverse Events
Description: An adverse event was any unfavorable and unintended sign, symptom, or disease associated with the use of the study drug, whether or not considered related to the study drug.
Time Frame: Up to 2.6 Years
Population: Safety Population included all participants who received study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Combigan® Ophthalmic Solution
Number analyzed (Participants) | 732
Percentage of participants | 6.56

2. Primary Outcome: Percentage of Participants With Overall Improvement From Baseline in Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. The study doctor classified the overall improvement of the IOP change from Baseline into 3 categories: Improvement (effective), No Change or Exacerbation (ineffective). The percentage of participants with Improvement is reported.
Time Frame: Baseline, Week 4
Population: Efficacy Population included all participants who received study drug for > 4 weeks and had overall assessment data available.
Measure: Number; unit: Percentage of participants
Arm/Group | Combigan® Ophthalmic Solution
Number analyzed (Participants) | 699
Percentage of participants | 85.69

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed for up to 2.6 years
Arm/Group | Combigan® Ophthalmic Solution
Serious Adverse Events (participants affected / at risk) | 0/732
Other Adverse Events (participants affected / at risk) | 0/732

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.